CLINICAL TRIAL: NCT07335926
Title: Tele-Pilates for Primary Dysmenorrhea: A Randomized Controlled Trial on Pain, Symptoms, and Trunk Endurance
Brief Title: Tele-Pilates for Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assoc. Prof., Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: hilalbuse1
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Primary Dysmenorrhea
Keywords: tele-pilates; menstrual pain; muscle endurance
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Pilates Group (Experimental): Participants received 16 synchronous tele-Pilates sessions over 8 weeks (twice per week). Exercises followed the APPI method including stretching, core strengthening, pelvic floor training, and breathing-focused control.
  Interventions: Other: Tele-Pilates Exercise program; Behavioral: standardized menstrual health education online
- Control Group (Active Comparator): Participants received standardized menstrual health education online but no exercise intervention.
  Interventions: Behavioral: standardized menstrual health education online

INTERVENTIONS:
Other: Tele-Pilates Exercise program — The intervention consisted of a synchronous, supervised tele-Pilates exercise program delivered via video conferencing platforms twice per week for 8 weeks. Each session lasted approximately 50 minutes and followed clinical Pilates principles based on the APPI method. The program emphasized core activation, diaphragmatic breathing, pelvic alignment, and trunk stabilization through progressively structured movements. Real-time feedback from a physiotherapist ensured correct execution, adaptation to individual capacity, and consistent adherence. The exercise protocol also incorporated components such as pelvic floor activation, transversus abdominis training, and guided relaxation.
  Arms: Tele-Pilates Group
Behavioral: standardized menstrual health education online — The education module consisted of two 45-minute interactive sessions conducted by a physiotherapist and covered the physiology of the menstrual cycle, pathophysiology of primary dysmenorrhea, common symptoms, and non-pharmacological management strategies. Content also included lifestyle modifications such as hydration, nutrition, physical activity, stress reduction techniques, and proper menstrual hygiene practices. Educational materials were adapted from current evidence-based guidelines and delivered using digital slides and discussion-based formats to promote participant engagement and understanding.

SUMMARY:
This randomized controlled trial investigates the effectiveness of a synchronized tele-Pilates program on menstrual pain, symptom severity, physical disability, and trunk muscle endurance in women with primary dysmenorrhea (PD). The intervention includes 16 supervised online Pilates sessions delivered over eight weeks.

DETAILED DESCRIPTION:
Primary dysmenorrhea is a prevalent gynecological condition characterized by painful menstruation. Exercise, particularly core stabilization and mind-body methods like Pilates, may improve both physical and psychological symptoms associated with PD. In this single-center RCT, 34 women aged 18-35 with PD were randomized to either a Tele-Pilates group or a control group. The Pilates group received supervised online sessions twice weekly for 8 weeks. Outcomes included pain severity (VAS), symptom burden (MSQ), functional impairment (FEMD), disability (Oswestry LBP Index), and trunk muscle endurance (McGill tests). Findings demonstrated significant improvements in the Pilates group across all domains.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-35 years
* Regular menstrual cycles (28±7 days)
* VAS ≥5 for menstrual pain
* Diagnosed with primary dysmenorrhea

Exclusion Criteria:

* Secondary dysmenorrhea (e.g., endometriosis, fibroids)
* Pregnancy or use of intrauterine devices
* Significant comorbidities (e.g., spondylolisthesis)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility is limited to individuals who self-identify as women, as primary dysmenorrhea is a condition specific to those with a female reproductive system.
Enrollment: 34 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Menstrual pain severity | Change from baseline to post-intervention (8 weeks)
  Menstrual pain severity was assessed using a 10 cm Visual Analog Scale, where participants marked the most intense pain experienced during their last menstrual cycle.

SECONDARY OUTCOMES:
Menstrual symptom severity (Menstrual Symptom Questionnaire total score) | Change from baseline to post-intervention (8 weeks)
  The Menstrual Symptom Questionnaire is a 24-item self-report measure assessing the severity of menstrual-related symptoms across emotional, physical, and pain domains; each item is rated on a 5-point Likert scale (1 = never to 5 = always), yielding a total score range of 24 to 120, where higher scores indicate worse symptom severity.
Functional and emotional burden (Functional and Emotional Measure of Dysmenorrhea total score) | Change from baseline to post-intervention (8 weeks)
  Functional and Emotional Measure of Dysmenorrhea (FEMD) is a 14-item self-report scale assessing the functional and emotional impact of dysmenorrhea, with each item rated on a 5-point Likert scale (1 = not at all similar to my situation to 5 = very similar to my situation), yielding a total score range of 14 to 70, where higher scores indicate greater functional and emotional impairment.
Trunk muscle endurance (McGill tests: flexor muscles) | Change from baseline to post-intervention (8 weeks)
  Endurance of trunk flexor muscles was measured using McGill's standardized core endurance test protocol, with duration recorded in seconds.
Trunk muscle endurance (McGill tests: extensor muscles) | Change from baseline to post-intervention (8 weeks)
  Endurance of trunk extensor muscles was measured using McGill's standardized core endurance test protocol, with duration recorded in seconds.
Trunk muscle endurance (McGill tests: lateral flexor muscles) | Change from baseline to post-intervention (8 weeks)
  Endurance of trunk lateral flexor muscles was measured using McGill's standardized core endurance test protocol, with duration recorded in seconds.
Disability due to low back pain (Oswestry Index) | Change from baseline to post-intervention (8 weeks)
  The Oswestry Disability Index was used to measure functional disability related to low back pain, commonly accompanied by dysmenorrhea, a 10-item scale. Each item is scored from 0 to 5, resulting in a total score range of 0 to 50, where higher scores indicate greater levels of disability and functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal DENİZOĞLU KÜLLİ, Principal Investigator — İSTANBUL ATLAS ÜNİVERSİTESİ
Locations (1):
- Atlas University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD).